CLINICAL TRIAL: NCT02482636
Title: Assessment of Post Booster Antibody Responses in UK Infants Given a Reduced Priming Schedule of Meningococcal Serogroup B and 13 Valent Pneumococcal Conjugate Vaccines
Brief Title: Baby Vaccine Study (Sched3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University College, London (Other); Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OVG2015/03
Record Dates: First submitted 2015-06-16; First posted 2015-06-26 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Infectious Diseases
Keywords: infant immunisations; vaccines; paediatric; pneumococcal; meningococcal
MeSH Terms: conditions — Communicable Diseases | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; 13-valent pneumococcal vaccine; Heptavalent Pneumococcal Conjugate Vaccine; Rotavirus Vaccines; RIX4414 vaccine; 4CMenB vaccine; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Group 1 will receive the following interventions:
  * DTaP/IPV/Hib vaccine IM 0.5ml at 2, 3 and 4 months
  * 13 valent pneumococcal conjugate vaccine (PCV13) IM 0.5ml at 2, 4 and 12 months
  * Rotavirus vaccine oral 1.5ml at 2 and 3 months
  * 4-component Meningococcal B (4CMenB) vaccine IM 0.5ml given at 2, 4 and 12 months
  * Meningococcal C/Hib vaccine IM 0.5ml at 12 months
  * Measles/Mumps/Rubella (MMR) vaccine IM 0.5ml at 13 months
  Interventions: Biological: DTaP/IPV/Hib vaccine; Biological: 13 valent Pneumococcal Conjugate Vaccine; Biological: Rotavirus vaccine; Biological: 4-component Meningococcal B vaccine; Biological: Meningococcal C/Hib vaccine (MenC/Hib vaccine); Biological: Measles/Mumps/Rubella Vaccine (MMR vaccine)
- Group 2 (Other): Group 2 will receive the following interventions:
  * DTaP/IPV/Hib vaccine IM 0.5ml at 2, 3 and 4 months
  * 13 valent pneumococcal conjugate vaccine (PCV13) IM 0.5ml at 3 and 12 months (instead of current routine schedule of 2,4 and 12 months)
  * Rotavirus vaccine oral 1.5ml at 2 and 3 months
  * 4-component Meningococcal B (4CMenB) vaccine IM 0.5ml given at 2, 4 and 12 months
  * Meningococcal C/Hib vaccine IM 0.5ml at 12 months
  * Measles/Mumps/Rubella (MMR) vaccine IM 0.5ml at 13 months
  Interventions: Biological: DTaP/IPV/Hib vaccine; Biological: 13 valent Pneumococcal Conjugate Vaccine; Biological: Rotavirus vaccine; Biological: 4-component Meningococcal B vaccine; Biological: Meningococcal C/Hib vaccine (MenC/Hib vaccine); Biological: Measles/Mumps/Rubella Vaccine (MMR vaccine)

INTERVENTIONS:
Biological: DTaP/IPV/Hib vaccine — Given at 2, 3 and 4 months to Group 1 and 2
  Other Names: Infanrix-IPV-Hib
Biological: 13 valent Pneumococcal Conjugate Vaccine — Given at 2,4 and 12 months in group 1, given at 3 and 12 months in group 2
  Other Names: PCV 13; Prevenar
Biological: Rotavirus vaccine — Given at 2 and 3 months to Group 1 and 2
  Other Names: Rotarix
Biological: 4-component Meningococcal B vaccine — Given at 2, 4 and 12 months to Group 1 and 2
  Other Names: Bexsero
Biological: Meningococcal C/Hib vaccine (MenC/Hib vaccine) — Given at 12 months to Group1 and 2
  Other Names: Menitorix
Biological: Measles/Mumps/Rubella Vaccine (MMR vaccine) — Given at 13 months to Groups 1 and 2
  Other Names: Priorix; MMR II

SUMMARY:
This multicentre, parallel group, block randomised clinical trial aims to investigate the post booster antibody response in UK infants given a reduced priming schedule of meningococcal serogroup B vaccine and 13 valent pneumococcal conjugate vaccine. It will provide information about how best to include the meningococcal B vaccine (likely to be introduced late 2015) into the routine immunisation schedule.

The UK Department of Health provides a routine vaccination schedule for children in the UK and are advised by the Joint Committee on Vaccination and Immunisation (JCVI). The Department of Health have announced that the meningococcal B vaccine (Bexsero) be introduced to the routine schedule as a 2+1 schedule. Cost effectiveness could also be improved by removing the current MenC conjugate vaccine dose given at 3 months of age. There is no published immunogenicity data for Bexsero when given at 2, 4 and 12 months of age (2+1 schedule) and with concomitant Infanrix/IPV/Hib which has now replaced Pediacel in the infant programme.

This change to the schedule would result in three injections at 2, 4 and 12 months, and given previous reluctance among parents for three injections at one visit, an option to reduce PCV13 to a 1+1 schedule (priming dose at 3 months and booster at 12 months) will be assessed in this study.

DETAILED DESCRIPTION:
The study's primary objective is to assess antibody response to the pneumococcal vaccine after the final infant vaccinations at approximately 13 months of age, and secondary objectives include antibody response following meningococcal B and C vaccines, tetanus, diphtheria and pertussis vaccines. In addition, the effect of maternal pertussis vaccination in pregnancy on infant immune response to vaccines, the prevalence of carriage of pneumococcal serotypes at 12 and 18 months of age and reactogenecity following each vaccine will be assessed.

200 healthy children who have not yet received their routine infant immunisations will be enrolled between 8 and 12 weeks old. Participants will be randomised into one of two groups with differing vaccine schedules. Children in both groups will receive their routine immunisations with the following changes: the addition of 3 doses of a meningococcal B vaccine at 2, 4 and 12 months and a meningococcal C vaccine at 12 months only (instead of a dose at 3 and 12 months). The 2 groups will differ by the number of doses of the 13-valent pneumococcal vaccine (PCV13); to be given either at 2, 4, and 12 months of age (as currently given in the routine schedule) or at 3 and 12 months of age.

Each participant will have 2 blood tests: at 5 and 13 months of age, and 2 nose swabs: at 12 and 18 months of age to address the objectives of the study. Parents will be asked to complete a health diary to record any adverse events in the 7 days following vaccinations and a continuous thermometer (ibutton) will be used to record the temperature for 24 hours after each vaccination.

If the blood samples at 13 months reveal antibody titres that are below the level indicative of protection, a recommendation will be made for booster vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Infants due to receive their primary immunisations , aged up to 13 weeks on first vaccinations.
* Written informed consent given by mother who is aged >= 16 years [NB mother is preferable as consent also allows permission to record the date of pertussis immunisation in pregnancy, which may need to be verified in her medical record. Where mother is not available, consent may be taken from father or legal guardian and maternal pertussis status noted as not known]

Exclusion Criteria:

* Bleeding disorder
* Fulfil any of the contraindications to vaccination as specified in The Green Book [https://www.gov.uk/government/organisations/public-health-england/series/immunisation-against-infectious-disease-the-green-book]:
* At risk of invasive pneumococcal disease (IPD) as defined in the Green Book pneumococcal chapter and those born prior to 37 weeks gestation
* Confirmed anaphylactic reaction to a previous dose of the vaccine, or
* Confirmed anaphylactic reaction to any constituent or excipient of the vaccine(s).
* A confirmed anaphylactic reaction to neomycin, streptomycin or polymyxin B (which may be present in trace amounts in the tetanus vaccine) and/or kanamycin, histidine, sodium chloride or sucrose (which may be present in trace amounts in the MenB vaccine).
* Latex hypersensitivity (the syringe cap of Bexsero may contain natural rubber latex)

Ages: 8 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 189 (Actual)
Dates: Start 2015-08; Primary Completion 2017-11-01 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Pneumococcal serotype specific geometric mean concentrations (GMCs) in blood samples following the completion of either a 2, 4 and 12 month schedule of PCV13 vaccination, or only 3 and 12 month PCV13 vaccination | Blood samples collected at 13 months of age
  pneumococcal IgG concentration for the 13 serotypes contained in the vaccine

SECONDARY OUTCOMES:
13 serotype-specific pneumococcal IgG GMCs and functional pneumococcal antibodies and proportions greater than or equal to ≥0.35µg/mL for each serotype in blood samples taken at 5 and 13 months | blood samples taken at 5 and 13 months
Titres and proportions of participants achieving antibody responses to MenB vaccination human Serum Bactericidal Antibody (SBA) titres ≥4 for the three main vaccine antigen target MenB strains, 5/99 (NadA), NZ98/254 (PorA) and 44/76-SL (fHbp) | Blood samples taken at 5 months
Meningococcal serogroup C human SBA geometric mean titres (GMTs) and proportion of infants ≥4 (5 month blood only); rabbit SBA titres (GMT) and proportion of infants with titres 8 and 128 (13 month blood only) | blood samples taken at 5 months and 13 months
Meningococcal serogroup W hSBA GMTs and proportion of infants with titre ≥4 at 5 and 13 months of age | blood samples taken at 5 and 13 months
GMC of anti-PRP IgG [Hib antigen] and proportion of infants with concentrations of > 0.15µg/mL and 1.0µg/mL in the blood samples taken at 5 and 13 months of age | Blood samples taken at 5 and 13 months of age
GMC of IgG to pertussis antigens (PT, PRN, FHA and FIM 2 and 3) in the blood samples taken at 5 months of age | Blood samples taken at 5 months of age
GMC of anti-tetanus toxoid IgG and proportions ≥0.1 IU/mL and ≥1.0 IU/mL in the blood samples taken at 5 months of age | Blood samples taken at 5 months of age
GMC of anti-diphtheria toxoid IgG and proportions ≥0.1IU/mL and ≥1.0 IU/mL in the blood samples taken at 5 months of age | blood samples taken at 5 months of age
Frequency of carriage of identified pneumococcal serotypes from the nasal swab collected prior to the booster vaccinations at 12 months of age and six months later | Nasal swab taken at 12 months and 18 months
Number of participants with local adverse events at injection site and temperature as recorded in the daily health diary for the week following vaccination and any systemic symptoms. Temperature also recorded and analysed from the iButton system | Measurements following vaccinations at 2, 3, 4, 12 and 13 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Snape, Principal Investigator — Oxford Vaccine Group, Chief Investigator
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Goldblatt D, Southern J, Andrews NJ, Burbidge P, Partington J, Roalfe L, Valente Pinto M, Thalasselis V, Plested E, Richardson H, Snape MD, Miller E. Pneumococcal conjugate vaccine 13 delivered as one primary and one booster dose (1 + 1) compared with two primary doses and a booster (2 + 1) in UK infants: a multicentre, parallel group randomised controlled trial. Lancet Infect Dis. 2018 Feb;18(2):171-179. doi: 10.1016/S1473-3099(17)30654-0. Epub 2017 Nov 22. PMID 29174323
- [Derived] Davis K, Valente Pinto M, Andrews NJ, Goldblatt D, Borrow R, Findlow H, Southern J, Partington J, Plested E, Patel S, Holland A, Matheson M, England A, Hallis B, Miller E, Snape MD. Immunogenicity of the UK group B meningococcal vaccine (4CMenB) schedule against groups B and C meningococcal strains (Sched3): outcomes of a multicentre, open-label, randomised controlled trial. Lancet Infect Dis. 2021 May;21(5):688-696. doi: 10.1016/S1473-3099(20)30600-9. Epub 2021 Jan 8. PMID 33428870
- [Derived] Valente Pinto M, Davis K, Andrews N, Goldblatt D, Borrow R, Southern J, Nordgren IK, Vipond C, Plested E, Miller E, Snape MD. Understanding the reactogenicity of 4CMenB vaccine: Comparison of a novel and conventional method of assessing post-immunisation fever and correlation with pre-release in vitro pyrogen testing. Vaccine. 2020 Nov 17;38(49):7834-7841. doi: 10.1016/j.vaccine.2020.10.023. Epub 2020 Oct 24. PMID 33109390